CLINICAL TRIAL: NCT03154008
Title: Neural Predictors of Response to Cognitive Behavioral Therapy for Adolescent Depression
Brief Title: Predictors of Response to Treatment for Depression
Acronym: PORT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: The Klingenstein Third Generation Foundation (Other)
Responsible Party: Principal Investigator, Autumn Kujawa, Assistant Professor, Vanderbilt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00007070
Record Dates: First submitted 2017-05-12; First posted 2017-05-15 (Actual); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Adolescent Depression; Depression
Keywords: reward; emotion regulation; electroencephalogram; event-related potentials; cognitive behavior therapy
MeSH Terms: conditions — Depression; Emotional Regulation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active Treatment (Experimental): Group cognitive behavioral therapy (CBT) for 8 weeks.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — Cognitive Behavioral Therapy will follow the Adolescent Coping with Depression Course (CWD; Clarke et al., 1999), an established 16-session group treatment protocol, and consist of behavioral activation, relaxation skills, cognitive therapy, social skills, problem solving, and relapse prevention.

SUMMARY:
The current study will examine neurophysiological, specifically event-related potential (ERP), measures of emotional processing as predictors of response to cognitive behavior therapy for adolescent depression.

DETAILED DESCRIPTION:
Neurophysiological measures (i.e., event-related potentials) of reward responsiveness and regulation of mood-congruent, sad stimuli will be assessed in a sample of adolescents with depression prior to group cognitive behavior therapy (CBT). CBT will follow the Adolescent Coping with Depression Course, an established 16-session group treatment protocol, and consist of behavioral activation, relaxation skills, cognitive therapy, social skills, problem solving, and relapse prevention. Changes in symptoms will be monitored through biweekly self-report and clinician ratings to examine prediction of change in symptoms across CBT. Baseline individual differences in reward responsiveness and emotion regulation will be evaluated as predictors of change in self-reported symptoms and clinician-rated improvement following CBT.

ELIGIBILITY:
Inclusion Criteria:

* Participants presenting with major depressive or persistent depressive disorder and moderate severity on the Clinical Global Impressions scale.
* Participants may have comorbid externalizing or anxiety disorders.
* Participants (and parents of minors) fluent in English.

Exclusion Criteria:

* Youth with history of treatment for substance use disorders.
* Youth with intellectual or developmental disabilities (e.g., autism spectrum disorders, pervasive developmental disorders).
* Youth with lifetime schizophrenia, psychosis, or mania.
* Youth with severe current suicidality.
* Youth taking antipsychotic medications or mood stabilizers.
* Youth with recent changes in dosage of antidepressant (adolescents with change in dosage in past 30 days who otherwise meet study criteria will be asked to begin the study once dosage has been stable for 30 days).
* Parent or child not fluent in English.
* Youth who are unable to complete study procedures because of visual or hearing impairments.
* Youth who have recently started outside therapy (past 30 days at time of intake), are engaged in treatment that is determined to be too similar to study therapy (e.g, other CBT groups), or are currently in treatment that is too intensive to allow for participation in study therapy (e.g., partial hospitalization programs)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2020-06-08 (Actual); Study Completion 2020-06-08 (Actual)

PRIMARY OUTCOMES:
Depressive symptoms | past 2 weeks
  Self-reported symptoms on the Mood and Feelings Questionnaire
Clinician-rated improvement | 8 weeks
  Global improvement rating on the Clinical Global Impression scale

CONTACTS AND LOCATIONS:
Overall Officials: Autumn Kujawa, PhD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Clarke GN, Rohde P, Lewinsohn PM, Hops H, Seeley JR. Cognitive-behavioral treatment of adolescent depression: efficacy of acute group treatment and booster sessions. J Am Acad Child Adolesc Psychiatry. 1999 Mar;38(3):272-9. doi: 10.1097/00004583-199903000-00014. PMID 10087688